CLINICAL TRIAL: NCT05594680
Title: The Phosphodiesterase 3 Inhibitor Cilostazol as Adjunct to Methotrexate in Patients With Rheumatoid Arthritis
Brief Title: Cilostazol and Methotrexate in Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Samar Mohammed Mahmoud Eldadamouny, Clinical Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: cilostazol in rheumatoid
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Cilostazol; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cilostazol and Methotrexate (Active Comparator): Participants in this arm will receive Cilostazol 50 mg twice daily with Methotrexate for rheumatoid arthritis for 12 weeks.
  Interventions: Drug: Cilostazol; Drug: Methotrexate
- Placebo and Methotrexate (Placebo Comparator): Participants in this arm will receive Placebo with Methotrexate for rheumatoid arthritis for 12 weeks.
  Interventions: Drug: Methotrexate; Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 50 MG
  Arms: Cilostazol and Methotrexate
Drug: Methotrexate — Methotrexate (MTX) is the first-line therapy for treatment of RA patients. MTX suppresses proliferation of synovial fibroblasts, modulates cytokine synthesis and superoxide anion production, and inhibits neutrophil chemotaxis.
Drug: Placebo — Placebo
  Arms: Placebo and Methotrexate

SUMMARY:
This study aims at evaluating the therapeutic effects of Cilostazol as adjuvant therapies to low dose of Methotrexate in patients with Rheumatoid Arthritis and to evaluate their impact on Cyclic adenosine monophosphate(CAMP), Heme Oxygenase-1(HO-1).

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is characterized by the presence of hyperplastic synovium in association with immune-mediated inflammatory synovitis associated with chronic production of proinflammatory cytokines, which lead to cartilage and bone degradation .This study is a randomized, controlled double blind placebo-controlled ,prospective study to evaluate the potential therapeutic effects of Cilostazol on synovial inflammation when administered as add-on treatments to the low dose of Methotrexate.

A total of 70 RA patients with active disease will be recruited from Outpatient Clinic of Physical Medicine, Rheumatology and Rehabilitation at Mansoura University hospitals, Mansoura, Egypt will be included in the study. They will be diagnosed with RA according to the American College of Rheumatology/European League Against Rheumatism criteria 2010 (the ACR/EULAR 2010 criteria).

RA Patients who will meet the inclusion criteria will be enrolled in the study.

They will be classified into two groups:

Group 1: 35 RA patients who will receive Methotrexate and placebo for 12 weeks and serve as the control group.

Group 2: 35 RA patients who will receive Methotrexate and Cilostazol 50 mg twice daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis (not in remission) according to American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2010 criteria (13) i.e 28 joints disease activity score (DAS-28) >2.6.
* Age range between 18 and 60 years old.
* Patients receive methotrexate; approximately the same doses of non steroidal anti-inflammatory drugs, selective cyclooxygenase-2 inhibitors, acetaminophen, and low dose of oral corticosteroids (Prednisolone < 15 mg) will be allowed to enroll the trial.
* Intravenous, intra-articular or intramuscular corticosteroids; intra articular hyaluronate sodium; biological DMARDs and other conventional DMARDs will not be permitted less than 4 weeks before the first dose of cilostazol.

Exclusion Criteria:

* Patients with diabetes, congestive heart failure, other heart disease (arrhythmia, hypertension, ischemic heart diseases), severe anemia, bleeding problems, other inflammatory diseases, active infection, other illness except rheumatoid arthritis.
* Patients on low doses of aspirin
* Patients on anticoagulants.
* Patients with renal or hepatic diseases.
* Patients receiving oral prednisolone greater than 15 mg/day.
* Patients receiving biological DMARDs.
* Patients with hypersensitivity to study medications.
* Patients using antioxidants .
* Pregnant and lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
change in DAS-28 CRP score | Baseline,12 weeks
  Clinical assessment by calculating of 28-joint count Disease Activity score (DAS-28) using C-reactive protein according to calculating formula(DAS28 (CRP) = 0.56*√(Tender joint count28) +0.28*√(Sowallen joint count28)+0.36*ln (CRP+1)*1.10+1.15 will done where high disease activity ≥ 5.1, low disease activity
  ≤ 3.2, and remission < 2.6.
Change in Multi Dimensional Health Assessment score | Baseline,12weeks
  Functional assessment will be assessed through Multi Dimensional Health Assessment score that include 14 items Health Assessment Questionaire .The score of the HAQ Questionnaire is calculated from the mean of the sum of the responses of the items where each item is scored from 0-3, where 0 = without any difficulty, 1
  = with some difficulty, 2 = with much difficulty, and 3 = unable to do. in addition, MDHAQ includes the assessment of morning stiffness (MS) duration in minutes.
Change in Visual analog scale for pain | Baseline,12 weeks
  Visual analog scales which ranges from 0 to 10,it is a psychometric scale that is generally used in hospitals and clinics by doctors to conduct pain scale surveys to understand varying degrees of pain or discomfort experienced by a patient.

SECONDARY OUTCOMES:
Change in the serum level of the assessed biological marker C-reactive protein | Baseline,12weeks
  C-reactive protein :CRP value (normal range <1.0 mg/dl). If the value is increased, the disease activity worsened. If the value is reduced the disease activity is improved.
Change in the serum level of the assessed biological marker Nuclear factor kabba-B p65 | Baseline,12weeks
  Transcriptional factor involved intracellular responses to stimuli and stress .So If the value is increased, the disease activity worsened. If the value is reduced the disease activity is improved.
Change in the serum level of the assessed biological marker Hemeoxygenase-1 | Baseline,12weeks
  Hemeoxygenase-1 .
Change in the serum level of the assessed biological marker Cyclic adenosine monophosphate | Baseline,12weeks
  Cyclic adenosine monophosphate level.

OTHER OUTCOMES:
Numbers of participants with treatment-related adverse events | Baseline,12weeks
  The adverse events in each group will be observed and documented during the whole procedure to show the safety of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Al Mansurah, Egypt

REFERENCES:
- [Background] Kim HY, Lee SW, Park SY, Baek SH, Lee CW, Hong KW, Kim CD. Efficacy of concurrent administration of cilostazol and methotrexate in rheumatoid arthritis: pharmacologic and clinical significance. Life Sci. 2012 Sep 17;91(7-8):250-7. doi: 10.1016/j.lfs.2012.07.003. Epub 2012 Jul 20. PMID 22820172
- [Background] Park SY, Lee SW, Kim HY, Lee SY, Lee WS, Hong KW, Kim CD. Suppression of RANKL-induced osteoclast differentiation by cilostazol via SIRT1-induced RANK inhibition. Biochim Biophys Acta. 2015 Oct;1852(10 Pt A):2137-44. doi: 10.1016/j.bbadis.2015.07.007. Epub 2015 Jul 11. PMID 26170060
- [Background] Kirino Y, Takeno M, Murakami S, Kobayashi M, Kobayashi H, Miura K, Ideguchi H, Ohno S, Ueda A, Ishigatsubo Y. Tumor necrosis factor alpha acceleration of inflammatory responses by down-regulating heme oxygenase 1 in human peripheral monocytes. Arthritis Rheum. 2007 Feb;56(2):464-75. doi: 10.1002/art.22370. PMID 17265482
- [Background] Park SY, Lee SW, Shin HK, Chung WT, Lee WS, Rhim BY, Hong KW, Kim CD. Cilostazol enhances apoptosis of synovial cells from rheumatoid arthritis patients with inhibition of cytokine formation via Nrf2-linked heme oxygenase 1 induction. Arthritis Rheum. 2010 Mar;62(3):732-41. doi: 10.1002/art.27291. PMID 20131233
- [Derived] Eldadamony SM, El-Haggar SM, Ali AMA, Mostafa TM. Clinical study evaluating the efficacy and safety of Cilostazol as an adjuvant therapy to methotrexate on patients with rheumatoid arthritis. Inflammopharmacology. 2025 Jun;33(6):3499-3508. doi: 10.1007/s10787-025-01782-2. Epub 2025 May 16. PMID 40380042